CLINICAL TRIAL: NCT01774864
Title: Phase 3 Study to Evaluate the Efficacy and Safety of Once-a-day Dosing of Udenafil in the Treatment of Erectile Dysfunction
Brief Title: Efficacy and Safety Study of Udenafil to Treat Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA8159_EDD_III
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DA-8159 dose 1 (Experimental): Udenafil
  Interventions: Drug: DA-8159 (Udenafil)
- DA-8159 dose 2 (Experimental): Udenafil
  Interventions: Drug: DA-8159 (Udenafil)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-8159 (Udenafil)
  Arms: DA-8159 dose 1; DA-8159 dose 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study Design : multi-center, double-blind, placebo-controlled, randomized,

parallel group, fixed dose design

Phase : Phase III

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 20 years or more diagnosed with ED

Exclusion Criteria:

* Had uncontrolled blood pressure
* Had hepatic or renal dysfunction
* Was currently under anticancer chemotherapy
* Had a treatments for ED using other PDE-5 inhibitors

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
IIEF EF domain score | 24 weeks

SECONDARY OUTCOMES:
IIEF, IPSS | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: S W Kim, MD, PhD, Principal Investigator — the Catholic University of Korea St. Mary's Hospital; D G Moon, MD, PhD, Principal Investigator — Korea University Guro Hospital; J J Kim, MD, PhD, Principal Investigator — Korea University Anam Hospital; N C Park, MD, PhD, Principal Investigator — Pusan National University Hospital; S W Lee, MD, PhD, Principal Investigator — Samsung Medical Center; J S Paick, MD, PhD, Principal Investigator — Seoul National University Hospital; T Y Ahn, MD, PhD, Principal Investigator — Asan Medical Center; K H Moon, MD, PhD, Principal Investigator — Yeungnam University Hospital; W S Chung, MD, PhD, Principal Investigator — Ewha Womans University; K S Min, MD, PhD, Principal Investigator — Inje University; J K Park, MD, PhD, Principal Investigator — Chonbuk National University Hospital; D Y Yang, MD, PhD, Principal Investigator — Kangdong Sacred Heart Hospital